CLINICAL TRIAL: NCT05843942
Title: Developing A Food Frequency Questionnaire To Evaluate Women's Dietary Iron, Folate, and Vitamin B12 Intake Status
Brief Title: Women's Health Food Frequency Questionnaire
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Zeynep Goktas, Principal Investigator, Hacettepe University
Other Study IDs: GO 22/867
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Diet Habit
Keywords: women's health; folate intake; iron intake; vitamin B12 intake
MeSH Terms: conditions — Feeding Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-pregnant women of reproductive age: In the first stage, a three-day food consumption record will be taken from 50 non-pregnant (menstruating) women of reproductive age in order to determine the foods to be included in the food consumption frequency section, and the questionnaire sections and questions (nutrition habits and food consumption frequency questionnaire) will be designed. In the second stage of the study, the questionnaire developed in the first stage will be applied to 350 non-pregnant (menstruating) volunteer women of reproductive age through face-to-face interviews. A 24-hour recall food consumption record will be taken. In this stage, the blood parameters of at least 100 individuals whose blood counts have already been taken for routine tests and treatments and who meet the inclusion criteria. In the third stage, the questionnaire will be applied again to 75 individuals who have completed the second stage at least 2 weeks later in order to evaluate the reliability of the questionnaire results.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — A food frequency questionnaire that was designed to assess folate, iron, and vitamin B12 intake will be administered. Furthermore a 24-hour recall food record will be administered and a complete blood count will be collected. Food frequency questionnaire data will be compared to recall food records and blood count data.

SUMMARY:
The aim of this study is to develop a tool that can measure the iron, folate, and vitamin B12 content of a diet through a literature review, database search, and a pilot study using a food consumption record. This tool will be used to accurately evaluate the iron, folate, and vitamin B12 content of the diet in non-pregnant women of reproductive age who are not currently pregnant. The research will be conducted on 350 women between the ages of 18 and 50 who are of reproductive age (menstruating). A questionnaire will be administered to the volunteer participants, which will consist of sections on general information, dietary habits, frequency of food consumption, and a 24-hour dietary recall.

DETAILED DESCRIPTION:
The study is planned in three stages. In the first stage, a three-day food consumption record will be taken from 50 non-pregnant (menstruating) women of reproductive age in order to determine the foods to be included in the food consumption frequency section, and the questionnaire sections and questions (nutrition habits and food consumption frequency questionnaire) will be designed. In the second stage of the study, the questionnaire developed in the first stage will be applied to 350 non-pregnant (menstruating) volunteer women of reproductive age through face-to-face interviews. In this stage, the blood parameters of at least 100 individuals whose blood counts have already been taken for routine tests and treatments and who meet the inclusion criteria of the study will also be recorded from their patient files. In the third stage, the questionnaire will be applied again to 75 individuals who have completed the second stage at least 2 weeks later in order to evaluate the reliability of the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* Between the ages of 19-50
* Of reproductive age
* Not pregnant
* Menstruating
* Not having a disease that affects nutrition
* Not following a special diet (weight loss diet, etc.)

Exclusion Criteria:

* Male sex
* Under 19 or over 50 years of age
* Having a disease that affects nutrition
* Following a special diet (gluten-free diet, etc.)
* Making changes in diet for the purpose of weight loss
* Of reproductive age but not menstruating

Ages: 19 Years to 50 Years | Sex: Female
Age Groups: Adult
Study Population: The sample of the study will consist of 350 non-pregnant (menstruating) volunteer women between the ages of 18-50 of reproductive age. The required sample size was calculated as 323 women via power analysis with a predicted 0.50 kappa agreement value, %5 type I error, and %95 confidence level. Subjects who meet the inclusion criteria of the study will be recruited among women that apply to the Hacettepe University Family Medicine Department Student Health Center.
Sampling Method: Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Iron intake | 12 months
  Dietary iron intake levels collected from both food frequency questionnaire and 24-hour recall food records
Folate intake | 12 months
  Dietary folate intake levels collected from both food frequency questionnaire and 24-hour recall food records
Vitamin B12 intake | 12 months
  Dietary vitamin B12 intake levels collected from both food frequency questionnaire and 24-hour recall food records

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Goktas, PhD, Principal Investigator — Hacettepe University
Locations (2):
- Turkey (Türkiye) (2):
  - Hacettepe University Family Medicine Department Student Health Center, Ankara
  - Hacettepe University Nutrition and Dietetics Department, Ankara

IPD SHARING:
Plan to Share IPD: No
The data are not publicly available due to privacy or ethical restrictions.